CLINICAL TRIAL: NCT01694485
Title: A Randomized, Double Blind, Multiple Dose Placebo Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of AMG 181 in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Abrilumab (AMG 181) in Adults With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110166; 2011-005251-13 (EudraCT Number)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis, IBD
MeSH Terms: conditions — Colitis, Ulcerative | interventions — abrilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo Q4W/Abrilumab 210 mg Q3M (Placebo Comparator): Participants received placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Biological: Abrilumab; Drug: Placebo
- Abrilumab 7 mg Q4W/Abrilumab 210 mg Q3M (Experimental): Participants received 7 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks (Q4W) thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Biological: Abrilumab
- Abrilumab 21 mg Q4W/Abrilumab 210 mg Q3M (Experimental): Participants received 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Biological: Abrilumab
- Abrilumab 70 mg Q4W/Abrilumab 210 mg Q3M (Experimental): Participants received 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Biological: Abrilumab
- Abrilumab 210 mg/Abrilumab 210 mg Q3M (Experimental): Participants received a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
  Interventions: Biological: Abrilumab; Drug: Placebo

INTERVENTIONS:
Biological: Abrilumab — Administered by subcutaneous injection.
  Other Names: AMG 181
Drug: Placebo — Placebo matching to abrilumab administered by subcutaneous injection
  Arms: Abrilumab 210 mg/Abrilumab 210 mg Q3M; Placebo Q4W/Abrilumab 210 mg Q3M

SUMMARY:
The primary objective of this study is to evaluate the effect of abrilumab on induction of remission in adults with moderate to severe ulcerative colitis after 8 weeks of treatment as assessed by a total Mayo Score ≤ 2 points, with no individual subscore > 1 point.

DETAILED DESCRIPTION:
The study consisted of a 24-week double-blind, placebo-controlled treatment period followed by an open-label period of approximately 108 weeks. Participants were eligible to enter the open-label period of the study early if they did not achieve a response at week 8 and had an inadequate response at week 12 or later or if they experienced disease worsening after achieving response and/or remission at week 8. Failure to achieve response at week 8 was defined as failure to achieve a decrease from baseline in total Mayo Score ≥ 3 points and ≥ 30% decrease from baseline. Inadequate response at week 12 or later was defined as failure to achieve a 2-point decrease and 25% improvement in partial Mayo Score compared with screening and minimum partial Mayo Score ≥ 5 points. Disease worsening was defined as an increase in partial Mayo Score ≥ 3 points from the week 8 value and minimum partial Mayo Score ≥ 5 points with recto-sigmoidoscopy sub-score ≥ 2.

Participants were planned to be randomized in a 2:1:2:2:2 ratio to placebo or abrilumab at 7 mg, 21 mg, 70 mg (on day 1, week 2, week 4, and every 4 weeks thereafter until week 24), or 210 mg (on day 1 followed by placebo in weeks 2 and 4 and every 4 weeks thereafter until week 24), respectively. Due to a consistent discrepancy between the investigational product (IP) instruction manual (IPIM) description of vial positions and the actual vial positions in the IP package participants were initially randomized to 3 arms (placebo, 70 mg, and 210 mg) with a randomization ratio of 4:3:2. The study was temporarily paused while this issue was investigated. Once the discrepancy was corrected, Protocol Amendment 3 implemented, and affected participants completed their double-blind treatment period, the study resumed enrollment and randomization per protocol. Neither the randomization nor study blind was compromised and therefore the intent-to-treat principle was maintained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis (UC) established ≥ 3 months before baseline by clinical and endoscopic evidence and corroborated by a histopathology report.
* Moderate to severe active UC as defined by a total Mayo score of 6 to 12 with a centrally read rectosigmoidoscopy score ≥2 prior to baseline
* Inadequate response to, loss of response to, or intolerance to at least one of the following treatments:

  * Immunomodulators
  * Anti-TNF agents
  * Corticosteroids (non-US sites only).
* Neurological exam free of clinically significant, unexplained signs or symptoms during screening and no clinically significant change prior to randomization

Exclusion Criteria:

* Disease limited to the rectum (ie, within 10 cm of the anal verge)
* Toxic megacolon
* Crohn's Disease
* History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for UC
* Planned bowel surgery within 24 weeks from baseline
* Stool positive for C. Difficile toxin at screening
* History of gastrointestinal surgery within 8 weeks of baseline
* Primary Sclerosing Cholangitis
* Any uncontrolled or clinically significant systemic disease
* Condition or disease that, in the opinion of the investigator would pose a risk to subject safety or interfere with study evaluation, procedures or completion.
* Known to have tested positive for hepatitis B virus surface antigen, hepatitis C virus antibody or human immunodeficiency virus (HIV)
* Underlying condition that predisposes subject to infections (eg, uncontrolled diabetes; history of splenectomy)
* Known history of drug or alcohol abuse within 1 year of screening
* Malignancy (other than resected cutaneous basal or cutaneous squamous cell carcinoma, or treated in situ cervical cancer considered cured) within 5 years of screening visit (if a malignancy occurred > 5 years ago, subject is eligible with documentation of disease free state since treatment)
* Immunosuppressive therapy with either cyclosporine A, tacrolimus, or mycophenolate mofetil, within 1 month prior to baseline
* Prior exposure to anti tumor necrosis factor (TNF) agents, within 2 months, or 5 times the respective elimination half life (whichever is longer) prior to baseline
* Any prior exposure to vedolizumab, rituximab, efalizumab, natalizumab
* Use of topical (rectal) aminosalicylic acid (eg, mesalamine) or topical (rectal) steroids within 2 weeks prior to baseline
* Use of intravenous or intramuscular corticosteroids within 2 weeks prior to screening and during screening
* Previously treated with AMG 181
* Received any type of live attenuated vaccine < 1 month prior to baseline or is planning to receive any such live attenuated vaccine over the course of the study
* Treatment of infection with intravenous (within 30 days of baseline) or oral (within 14 days prior to baseline) antibiotics, antivirals, or antifungals
* Abnormal laboratory results at screening
* Any other laboratory abnormality, which, in the opinion of the investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (112):
- United States (24):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, La Jolla, California
  - Research Site, Torrance, California
  - Research Site, Lone Tree, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Arlington Heights, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Hammond, Louisiana
  - Research Site, Chesterfield, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Mentor, Ohio
  - Research Site, Germantown, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Seattle, Washington
- Australia (4):
  - Research Site, Bankstown, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, Box Hill, Victoria
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Sankt Veit an der Glan
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Herlev
  - Research Site, Hvidovre
  - Research Site, Køge
  - Research Site, Odense C
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (8):
  - Research Site, Amiens
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (5):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, Kiel
- Greece (5):
  - Research Site, Athens
  - Research Site, Haidari
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Piraeus
- Hungary (7):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szekszárd
- Italy (6):
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano MI
- Research Site, Riga, Latvia
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Leiden
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Norway (2):
  - Research Site, Oslo
  - Research Site, Tromsø
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (6):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, St.-Petrsburg
  - Research Site, Stavropol
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Zurich
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Coventry
  - Research Site, Derby
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Norwich

REFERENCES:
- [Derived] Sandborn WJ, Cyrille M, Hansen MB, Feagan BG, Loftus EV Jr, Rogler G, Vermeire S, Cruz ML, Yang J, Boedigheimer MJ, Abuqayyas L, Evangelista CM, Sullivan BA, Reinisch W. Efficacy and Safety of Abrilumab in a Randomized, Placebo-Controlled Trial for Moderate-to-Severe Ulcerative Colitis. Gastroenterology. 2019 Mar;156(4):946-957.e18. doi: 10.1053/j.gastro.2018.11.035. Epub 2018 Nov 23. PMID 30472236
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 92 centers located in North America, Europe, and Australia from 16 November 2012 to 11 May 2015.
  The study consisted of a 24-week double-blind treatment period, a 108-week open-label treatment period, and a safety follow-up period.
Pre-assignment Details: Participants were to be randomly assigned in a 2:1:2:2:2 ratio to 1 of 5 treatment groups. Due to a misalignment error, some participants were erroneously assigned to incorrect treatment resulting in a final randomization ratio different from that originally stipulated in the protocol.
Groups:
- Placebo/Abrilumab 210 mg Q3M: Participants randomized to receive placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks.
- Abrilumab 7 mg Q4W/Abrilumab 210 mg Q3M: Participants randomized to receive 7 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks (Q4W) thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
- Abrilumab 21 mg Q4W/Abrilumab 210 mg Q3M: Participants randomized to receive 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
- Abrilumab 70 mg Q4W/Abrilumab 210 mg Q3M: Participants randomized to receive 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
- Abrilumab 210 mg/Abrilumab 210 mg Q3M: Participants randomized to receive a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24.
  During the open-label period, participants received abrilumab 210 mg once every 3 months for 108 weeks.
Period: Overall Study
Arm/Group | Placebo/Abrilumab 210 mg Q3M | Abrilumab 7 mg Q4W/Abrilumab 210 mg Q3M | Abrilumab 21 mg Q4W/Abrilumab 210 mg Q3M | Abrilumab 70 mg Q4W/Abrilumab 210 mg Q3M | Abrilumab 210 mg/Abrilumab 210 mg Q3M
Started | 117 | 22 | 40 | 100 | 80
Received Treatment | 116 | 21 | 40 | 98 | 79
Completed Week 8 Assessment | 106 | 18 | 38 | 94 | 76
Entered Open-label Period | 100 | 19 | 36 | 88 | 68
Completed (Defined as participants who completed the safety follow-up period) | 84 | 15 | 27 | 62 | 55
Not Completed | 33 | 7 | 13 | 38 | 25
Not completed — Withdrawal by Subject | 20 | 6 | 7 | 25 | 18
Not completed — Sponsor Decision | 3 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 9 | 1 | 6 | 10 | 7
Not completed — Death | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to receive placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Abrilumab 7 mg Q4W: Participants randomized to receive 7 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Abrilumab 21 mg Q4W: Participants randomized to receive 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Abrilumab 70 mg Q4W: Participants randomized to receive 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Abrilumab 210 mg: Participants randomized to receive a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Abrilumab 7 mg Q4W | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg | Total
Number analyzed (Participants) | 117 | 22 | 40 | 100 | 80 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.3) | 42.0 (12.4) | 38.3 (11.6) | 39.3 (12.2) | 39.8 (12.0) | 40.0 (12.5)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 113 | 22 | 40 | 99 | 80 | 354
  ≥ 65 years | 4 | 0 | 0 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 8 | 12 | 32 | 32 | 120
  Male | 81 | 14 | 28 | 68 | 48 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 2 | 0 | 3 | 9
  Not Hispanic or Latino | 113 | 22 | 38 | 100 | 77 | 350
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 2 | 1 | 7 | 1 | 16
  White | 109 | 20 | 39 | 89 | 78 | 335
  Other | 3 | 0 | 0 | 4 | 1 | 8
Any Prior Anti-Tumor Necrosis Factor (TNF) Use [Count of Participants; unit: Participants]
  Yes | 69 | 6 | 10 | 56 | 39 | 180
  No | 48 | 16 | 30 | 44 | 41 | 179
Enrollment Prior to Protocol Amendment 3 [Count of Participants; unit: Participants]
  Yes | 76 | 0 | 0 | 58 | 38 | 172
  No | 41 | 22 | 40 | 42 | 42 | 187
Duration of Ulcerative Colitis [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 116 | 22 | 40 | 100 | 80 | 358
    (all) | 7.83 (5.58) | 9.07 (6.57) | 7.05 (5.39) | 9.39 (7.25) | 9.44 (7.88) | 8.62 (6.70)
Total Mayo Score [Mean (Standard Deviation); unit: units on a scale] — The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a score of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  units on a scale | 8.9 (1.5) | 8.1 (1.4) | 8.6 (1.7) | 9.0 (1.5) | 9.1 (1.4) | 8.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission at Week 8
Description: Remission was defined as a total Mayo Score ≤ 2 points, with no individual subscore > 1 point.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a score of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  The remission rate (percentage of participants with remission) was calculated based on observed data (unadjusted remission rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline total Mayo Score (adjusted remission rate).
Time Frame: Week 8
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted remission rates were calculated using non-responder imputation, where participants with a missing Mayo Score at week 8 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 7 mg Q4W | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 116 | 21 | 40 | 98 | 79
percentage of participants
  Unadjusted remission rate | 4.3 | 0.0 | 2.5 | 13.3 | 12.7
  Adjusted remission rate | 4.4 | 1.6 | 2.9 | 13.5 | 13.4
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using remission rates estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — The study was powered for formal statistical testing of the abrilumab 70 mg and 210 mg groups. To account for multiplicity of statistical testing, primary and key secondary end points for the 2 highest doses of abrilumab (70 and 210 mg) were tested at the end of the 8-week induction period under a sequential framework at a 2-sided significance level of 0.10 using the Bonferroni-based chain procedure; p = 0.021, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 3.35, 90% CI 2-sided [1.41 to 7.95] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in remission rates, estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Remission Rates = 9.0, 90% CI 2-sided [1.6 to 14.6]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; Comparisons between treatment groups were made using remission rates from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.030, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 3.33, 90% CI 2-sided [1.34 to 8.26] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Difference in Adjusted Remission Rates = 8.9, 90% CI 2-sided [0.8 to 14.9]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Comparisons of abrilumab 21 mg with placebo were not included in the hypothesis testing procedure and were not adjusted for multiplicity; p = 0.64, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 0.64, 90% CI 2-sided [0.13 to 3.17] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; The difference in remission rates estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = -1.6, 90% CI 2-sided [-5.2 to 5.5]
Statistical Analysis 7: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 1, analysis 3]; Test type: Superiority — Comparisons of abrilumab 7 mg with placebo were not included in the hypothesis testing procedure and were not adjusted for multiplicity; p = 0.49, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 0.34, 90% CI 2-sided [0.03 to 4.33] — An odds ratio > 1.0 indicates a higher remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 8: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 1, analysis 6]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = -2.9, 90% CI 2-sided [-5.5 to 5.4]

2. Secondary Outcome: Percentage of Participants With Response at Week 8
Description: Response was defined by a decrease from baseline in the total Mayo Score of ≥ 3 points and ≥ 30%, with an accompanying decrease in the rectal bleeding subscore ≥ 1 point or an absolute rectal bleeding subscore = 0 or 1.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment), each graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, ranging from 0 to 12 points. Higher scores represent more severe disease.
  The response rate (percentage of participants with response) was calculated based on observed data (unadjusted response rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline total Mayo Score (adjusted response rate).
Time Frame: Baseline and week 8
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted response rates were calculated using non-responder imputation, where participants with a missing Mayo Score at week 8 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 7 mg Q4W | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 116 | 21 | 40 | 98 | 79
percentage of participants
  Unadjusted response rate | 25.9 | 14.3 | 50.0 | 49.0 | 46.8
  Adjusted response rate | 26.0 | 12.3 | 47.2 | 49.4 | 47.4
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using response rates estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — If both comparisons of the primary endpoint reached statistical significance at 0.10, results from the 2 key secondary endpoints (response and mucosal healing at week 8) were to be sequentially (70 mg vs placebo then 210 mg vs placebo) tested at significance level of 0.05 independently of each other, according to the Bonferroni-based chain procedure; p < 0.001, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 2.78, 90% CI 2-sided [1.71 to 4.52] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in adjusted response rates, estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Response Rates = 23.4, 90% CI 2-sided [11.8 to 33.2]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; Comparisons between treatment groups were made using response rates from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.003, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 2.57, 90% CI 2-sided [1.53 to 4.31] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Difference in Adjusted Response Rates = 21.4, 90% CI 2-sided [9.0 to 31.8]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 2, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 5]; p = 0.024, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 2.54, 90% CI 2-sided [1.29 to 5.02] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Response Rates = 21.2, 90% CI 2-sided [4.9 to 34.1]
Statistical Analysis 7: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 2, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.18, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 0.40, 90% CI 2-sided [0.13 to 1.22] — An odds ratio > 1.0 indicates a higher response rate for the abrilumab treatment group relative to placebo
Statistical Analysis 8: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 2, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Response Rates = -13.7, 90% CI 2-sided [-24.4 to 2.7]

3. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 8
Description: Mucosal healing was defined using the rectosigmoidoscopy subscore of Mayo assessment as absolute subscore for rectosigmoidoscopy of 0 or 1.
  Flexible rectosigmoidoscopy was performed as part of the Mayo assessment, graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status.
  The healing rate (percentage of participants with mucosal healing) was calculated based on observed data (unadjusted healing rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline rectosigmoidoscopy score (adjusted healing rate).
Time Frame: Week 8
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both unadjusted and adjusted healing rates were calculated using non-responder imputation, where participants with missing rectosigmoidoscopy scores at week 8 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 7 mg Q4W | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 116 | 21 | 40 | 98 | 79
percentage of participants
  Unadjusted healing rate | 21.6 | 14.3 | 15.0 | 32.7 | 29.1
  Adjusted healing rate | 16.8 | 12.2 | 13.9 | 32.2 | 29.8
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using healing rates estimated from a logistic regression model adjusted for baseline rectosigmoidoscopy score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.011, Regression, Logistic; Adjusted for baseline rectosigmoidoscopy score and stratification factors; Odds Ratio (OR) = 2.34, 90% CI 2-sided [1.35 to 4.07] — An odds ratio > 1.0 indicates a higher healing rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in adjusted healing rates, estimated from a logistic regression model adjusted for baseline rectosigmoidoscopy score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Healing Rates = 15.3, 90% CI 2-sided [4.8 to 24.0]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; Comparisons between treatment groups were made using healing rates from a logistic regression model adjusted for baseline rectosigmoidoscopy score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.041, Regression, Logistic; Adjusted for baseline rectosigmoidoscopy score and stratification factors; Odds Ratio (OR) = 2.10, 90% CI 2-sided [1.15 to 3.82] — An odds ratio > 1.0 indicates a higher healing rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; Difference in Adjusted Healing Rates = 13.0, 90% CI 2-sided [1.7 to 22.1]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 3, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 5]; p = 0.68, Regression, Logistic; Adjusted for baseline rectosigmoidoscopy score and stratification factors; Odds Ratio (OR) = 0.80, 90% CI 2-sided [0.32 to 1.97] — An odds ratio > 1.0 indicates a higher healing rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Healing Rates = -3.0, 90% CI 2-sided [-11.9 to 9.4]
Statistical Analysis 7: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 3, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.60, Regression, Logistic; Adjusted for baseline rectosigmoidoscopy score and stratification factors; Odds Ratio (OR) = 0.69, 90% CI 2-sided [0.21 to 2.22] — An odds ratio > 1.0 indicates a higher healing rate for the abrilumab treatment group relative to placebo
Statistical Analysis 8: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Healing Rates = -4.6, 90% CI 2-sided [-14.9 to 11.3]

4. Secondary Outcome: Percentage of Participants With Sustained Remission at Week 8 and Week 24
Description: Remission was defined as a total Mayo Score ≤ 2 points, with no individual subscore > 1 point. Sustained remission was defined as achieving the criteria for remission at both week 8 and week 24.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment), each graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher scores represent more severe disease status. The total Mayo Score is the sum of the four item scores, with a and ranges from 0 to 12 points. Higher scores represent more severe disease.
  The remission rate (percentage of participants with sustained remission) was calculated based on observed data (unadjusted remission rate) and also after applying a logistic regression model including the factors of treatment group, stratification factors (prior anti-TNF use and pre- versus post-Protocol Amendment 3) and baseline total Mayo Score (adjusted remission rate).
Time Frame: Week 8 and week 24
Population: The full analysis set includes all randomized participants who received at least 1 dose of study drug. Both non-adjusted and adjusted remission rates were calculated using non-responder imputation, where participants with missing Mayo Score at week 8 or week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Abrilumab 7 mg Q4W | Abrilumab 21 mg Q4W | Abrilumab 70 mg Q4W | Abrilumab 210 mg
Number analyzed (Participants) | 116 | 21 | 40 | 98 | 79
percentage of participants
  Unadjusted remission rate | 2.6 | 0.0 | 2.5 | 8.2 | 3.8
  Adjusted remission rate | 3.3 | 1.6 | 2.8 | 9.1 | 4.3
Statistical Analysis 1: Comparison: Placebo vs Abrilumab 70 mg Q4W; Comparisons between treatment groups were made using sustained remission rates estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; p = 0.090, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 2.94, 90% CI 2-sided [1.03 to 8.36] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 2: Comparison: Placebo vs Abrilumab 70 mg Q4W; The difference in adjusted sustained remission rates, estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; Difference in Adjusted Remission Rates = 5.8, 90% CI 2-sided [-0.6 to 10.4]
Statistical Analysis 3: Comparison: Placebo vs Abrilumab 210 mg; Comparisons between treatment groups were made using sustained remission rates from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority; p = 0.72, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 1.32, 90% CI 2-sided [0.38 to 4.56] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 4: Comparison: Placebo vs Abrilumab 210 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; Difference in Adjusted Remission Rates = 1.0, 90% CI 2-sided [-4.7 to 4.6]
Statistical Analysis 5: Comparison: Placebo vs Abrilumab 21 mg Q4W; [analysis description as in outcome 4, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 5]; p = 0.86, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 0.83, 90% CI 2-sided [0.16 to 4.41] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 6: Comparison: Placebo vs Abrilumab 21 mg Q4W; The difference in adjusted sustained remission rates estimated from a logistic regression model adjusted for baseline total Mayo Score and stratification factors (prior vs no prior TNF antagonist use and enrollment pre- vs post-protocol amendment); Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = -0.5, 90% CI 2-sided [-3.9 to 6.2]
Statistical Analysis 7: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 4, analysis 3]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.64, Regression, Logistic; Adjusted for baseline total Mayo Score and stratification factors; Odds Ratio (OR) = 0.49, 90% CI 2-sided [0.04 to 6.31] — An odds ratio > 1.0 indicates a higher sustained remission rate for the abrilumab treatment group relative to placebo
Statistical Analysis 8: Comparison: Placebo vs Abrilumab 7 mg Q4W; [analysis description as in outcome 4, analysis 6]; Test type: Superiority — Analysis was not part of the formal testing; Difference in Adjusted Remission Rates = -1.7, 90% CI 2-sided [-4.2 to 6.4]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to week 24 in the double-blind period and from first dose of study drug in the open-label period to 12 weeks after last dose in the open-label period (up to 108 weeks).
Description: One participant who was randomized to the 7 mg abrilumab arm was treated with 70 mg abrilumab and is counted in the Abrilumab 70 mg group for safety assessments in both treatment periods.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- DB Period: Placebo: Participants received placebo by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind (DB) treatment period.
- DB Period: Abrilumab 7 mg Q4W: Participants received 7 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks (Q4W) thereafter until week 24 during the double-blind treatment period.
- DB Period: Abrilumab 21 mg Q4W: Participants received 21 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- DB Period: Abrilumab 70 mg Q4W: Participants received 70 mg abrilumab by subcutaneous injection on day 1, week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- DB Period: Abrilumab 210 mg: Participants received a single dose of 210 mg abrilumab by subcutaneous injection on day 1, followed by placebo at week 2, week 4, and every 4 weeks thereafter until week 24 during the double-blind treatment period.
- OL Period: Placebo/Abrilumab 210 mg Q3M: Participants who received placebo during the double-blind treatment period received abrilumab 210 mg once every 3 months (Q3M) for 108 weeks during the open-label (OL) treatment period.
- OL Period: Abrilumab 7 mg Q4W/210 mg Q3M: Participants who received 7 mg abrilumab Q4W in the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks during the open-label period.
- OL Period: Abrilumab 21 mg Q4W/210 mg Q3M: During the open-label period, participants who received 21 mg abrilumab Q4W during the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks.
- OL Period: Abrilumab 70 mg Q4W/210 mg Q3M: Participants who received 70 mg abrilumab Q4W during the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks during the open-label period.
- OL Period: Abrilumab 210 mg/210 mg Q3M: Participants who received 210 mg abrilumab during the DB treatment period received abrilumab 210 mg once every 3 months for 108 weeks during the open-label period.
Arm/Group | DB Period: Placebo | DB Period: Abrilumab 7 mg Q4W | DB Period: Abrilumab 21 mg Q4W | DB Period: Abrilumab 70 mg Q4W | DB Period: Abrilumab 210 mg | OL Period: Placebo/Abrilumab 210 mg Q3M | OL Period: Abrilumab 7 mg Q4W/210 mg Q3M | OL Period: Abrilumab 21 mg Q4W/210 mg Q3M | OL Period: Abrilumab 70 mg Q4W/210 mg Q3M | OL Period: Abrilumab 210 mg/210 mg Q3M
Serious Adverse Events (participants affected / at risk) | 14/116 | 1/20 | 3/40 | 5/99 | 7/79 | 13/100 | 3/18 | 4/36 | 14/89 | 6/68
Other Adverse Events (participants affected / at risk) | 47/116 | 9/20 | 16/40 | 55/99 | 35/79 | 55/100 | 10/18 | 19/36 | 53/89 | 26/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=116) | DB Period: Abrilumab 7 mg Q4W (N=20) | DB Period: Abrilumab 21 mg Q4W (N=40) | DB Period: Abrilumab 70 mg Q4W (N=99) | DB Period: Abrilumab 210 mg (N=79) | OL Period: Placebo/Abrilumab 210 mg Q3M (N=100) | OL Period: Abrilumab 7 mg Q4W/210 mg Q3M (N=18) | OL Period: Abrilumab 21 mg Q4W/210 mg Q3M (N=36) | OL Period: Abrilumab 70 mg Q4W/210 mg Q3M (N=89) | OL Period: Abrilumab 210 mg/210 mg Q3M (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 5 | 0 | 1 | 4 | 2 | 6 | 0 | 2 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Norovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=116) | DB Period: Abrilumab 7 mg Q4W (N=20) | DB Period: Abrilumab 21 mg Q4W (N=40) | DB Period: Abrilumab 70 mg Q4W (N=99) | DB Period: Abrilumab 210 mg (N=79) | OL Period: Placebo/Abrilumab 210 mg Q3M (N=100) | OL Period: Abrilumab 7 mg Q4W/210 mg Q3M (N=18) | OL Period: Abrilumab 21 mg Q4W/210 mg Q3M (N=36) | OL Period: Abrilumab 70 mg Q4W/210 mg Q3M (N=89) | OL Period: Abrilumab 210 mg/210 mg Q3M (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 2 | 4 | 1 | 3 | 6 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 1 | 8 | 1 | 3 | 6 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 4 | 0 | 2 | 7 | 6 | 17 | 4 | 11 | 22 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 5 | 2 | 0 | 2 | 5 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 4 | 5 | 2 | 1 | 1 | 5 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 2 | 4 | 1 | 2 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 4 | 1
Fatigue (General disorders) | 3 | 0 | 1 | 8 | 3 | 1 | 0 | 1 | 1 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 4 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 4 | 0 | 2 | 0 | 3 | 3 | 1
Influenza (Infections and infestations) | 4 | 2 | 0 | 2 | 0 | 3 | 1 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 7 | 0 | 6 | 9 | 8 | 9 | 0 | 1 | 5 | 6
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 4 | 1 | 5 | 0 | 2 | 5 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 4 | 11 | 6 | 11 | 2 | 3 | 9 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 2 | 1 | 5 | 0 | 0 | 8 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 1 | 2 | 11 | 8 | 3 | 2 | 1 | 5 | 4
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5 | 2 | 2 | 0 | 1 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 3 | 3 | 1 | 0 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 4 | 1 | 5 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.